CLINICAL TRIAL: NCT00666705
Title: An Open Label Phase 4 Study To Evaluate An Interaction Between Maraviroc And Raltegravir In Healthy Subjects
Brief Title: A Study To Evaluate An Interaction Between Maraviroc And Raltegravir In Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: A4001082
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Results first posted 2009-06-04 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: maraviroc; raltegravir; drug interaction study; healthy volunteers
MeSH Terms: interventions — Maraviroc; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Maraviroc alone (Experimental)
  Interventions: Drug: Maraviroc
- Maraviroc + Raltegravir (Experimental)
  Interventions: Drug: Maraviroc; Drug: Raltegravir
- Raltegravir alone (Experimental)
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Maraviroc — 300 milligrams(mg) every 12 hours Days 6-11
  Other Names: Selzentry, Celsentri
  Arms: Maraviroc alone
Drug: Maraviroc — Days 12-14: Raltegravir 400 milligrams(mg) every 12 hours, maraviroc 300 milligrams(mg) every 12 hours (AM doses only on Day 14)
  Arms: Maraviroc + Raltegravir
Drug: Raltegravir — Days 12-14: Raltegravir 400 milligrams(mg) every 12 hours, maraviroc 300 milligrams(mg) every 12 hours (AM doses only on Day 14)
  Arms: Maraviroc + Raltegravir
Drug: Raltegravir — 400 milligrams(mg) every 12 hours Days 1-3 Followed by washout Days 4-5
  Arms: Raltegravir alone

SUMMARY:
An open label study to evaluate an interaction between maraviroc and raltegravir in healthy subjects.

DETAILED DESCRIPTION:
Drug interaction study

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between 18 and 55 years of age.

Exclusion Criteria:

* Evidence or history of clinically significant disease or clinical findings at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001082&StudyName=A%20Study%20To%20Evaluate%20An%20Interaction%20Between%20Maraviroc%20And%20Raltegravir%20In%20Healthy%20Subjects

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One site in the United States
Pre-assignment Details: Subjects were to be healthy male or female subjects between the ages of 18 and 55 years, inclusive. Subjects were required to meet all eligibility criteria prior to randomization into the study.
Groups:
- Maraviroc / Raltegravir (Alone and Co-administered): All subjects received the following fixed sequence study treatments:
  Days 1-3: raltegravir 400 milligrams (mg) every 12 hours (AM dose on Day 3) Days 4-5: washout Days 6-11: maraviroc 300 mg every 12 hours Days 12-14: raltegravir 400 mg every 12 hours and maraviroc 300 mg every 12 hours (AM doses on Day 14).
Period: Overall Study
Arm/Group | Maraviroc / Raltegravir (Alone and Co-administered)
Started | 18
Raltegravir Alone (Days 1 - 3) | 18 (400 mg Raltegravir every 12 hours (AM dose on Day 3))
Washout (Days 4 - 5) | 18
Maraviroc Alone (Days 6 - 11) | 18 (300 mg Maraviroc every 12 hours)
Raltegravir + Maraviroc (Days 12 - 14) | 17 (400 mg Raltegravir every 12 hours plus 300 mg Maraviroc every 12 hours (AM doses only on Day 14))
Completed | 17
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Maraviroc / Raltegravir (Alone and Co-administered): All subjects received the following fixed sequence study treatments:
  Days 1-3: raltegravir 400 mg every 12 hours (AM dose on Day 3) Days 4-5: washout Days 6-11: maraviroc 300 mg every 12 hours Days 12-14: raltegravir 400 mg every 12 hours and maraviroc 300 mg every 12 hours (AM doses on Day 14).
Arm/Group | Maraviroc / Raltegravir (Alone and Co-administered)
Number analyzed (Participants) | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 36.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Maraviroc Pharmacokinetic (PK) Parameter: Area Under the Plasma Concentration-time Profile Over the Dosing Interval (AUCτ)
Description: Effect of raltegravir on pharmacokinetics of maraviroc (comparison of AUCτ of raltegravir co-administered with maraviroc (Test) versus maraviroc administered alone (Reference)). Pharmacokinetics were assessed on Day 11 (maraviroc) and Day 14 (maraviroc and raltegravir).
Time Frame: Days 11 and 14
Population: The Pharmacokinetic (PK) parameter analysis population is defined as all subjects enrolled and treated who have at least one of the PK parameters of primary interest in at least one treatment period.
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Groups:
- Maraviroc + Raltegravir (Test): On Study Days 12-14: Raltegravir 400 mg every 12 hours, maraviroc 300 mg every 12 hours (AM doses only on Day 14)
- Maraviroc (Reference): 300 mg every 12 hours on Study Days 6-11
Arm/Group | Maraviroc + Raltegravir (Test) | Maraviroc (Reference)
Number analyzed (Participants) | 17 | 17
ng.hr/mL | 2551.9 (786.68) | 2971.6 (841.65)
Statistical Analysis 1: Comparison: Maraviroc + Raltegravir (Test) vs Maraviroc (Reference); The alternate hypothesis of bioequivalence is that there is no difference between treatment groups. For maraviroc, a sample size of 18 subjects provided 99% power that the 90% confidence interval (CI) for the ratio of Test (raltegravir co-administered with maraviroc) to Reference (maraviroc administered alone) treatment for the area under the plasma concentration-time profile over the dosing interval (AUCτ) would lie within the acceptance region of (80%, 125%); Test type: Superiority or Other; Mixed Models Analysis; Natural log transformed AUCτ was analyzed using a mixed effect model with treatment as a fixed effect and subject as a random effect; Ratio (percent) = 85.76, 90% CI [79.89 to 92.07] — Ratio (percent) (Test/Reference) of Adjusted Geometric Means

2. Primary Outcome: Maraviroc Pharmacokinetic (PK) Parameter: Maximum Concentration (Cmax)
Description: Effect of raltegravir on pharmacokinetics of maraviroc (comparison of Cmax of raltegravir co-administered with maraviroc (Test) versus maraviroc administered alone (Reference)). Pharmacokinetics were assessed on Day 11 (maraviroc) and Day 14 (maraviroc and raltegravir). Cmax is the maximum plasma concentration.
Time Frame: Days 11 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Maraviroc + Raltegravir (Test) | Maraviroc (Reference)
Number analyzed (Participants) | 17 | 17
ng/mL | 691.6 (322.24) | 851.4 (349.38)
Statistical Analysis 1: Comparison: Maraviroc + Raltegravir (Test) vs Maraviroc (Reference); The alternate hypothesis of bioequivalence is that there is no difference between treatment groups. For maraviroc, a sample size of 18 subjects provided 91% power that the 90% CI for the ratio of Test (raltegravir co-administered with maraviroc) to Reference (maraviroc administered alone) treatment for the maximum concentration (Cmax) would lie within the acceptance region of (80%, 125%); Test type: Superiority or Other; Mixed Models Analysis; Natural log transformed Cmax was analyzed using a mixed effect model with treatment as a fixed effect and subject as a random effect; Ratio (percent) = 79.48, 90% CI [67.19 to 94.02] — Ratio (percent) (Test/Reference) of Adjusted Geometric Means

3. Primary Outcome: Raltegravir Pharmacokinetics (PK) Parameter: Area Under the Plasma Concentration-time Profile Over the Dosing Interval (AUCτ)
Description: Effect of maraviroc on pharmacokinetics of raltegravir (comparison of AUCτ of raltegravir co-administered with maraviroc (Test) versus raltegravir administered alone (Reference)). Pharmacokinetics were assessed on Day 3 (raltegravir) and Day 14 (maraviroc and raltegravir).
Time Frame: Days 3 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Groups:
- Maraviroc + Raltegravir (Test): On Study Days 12-14: Raltegravir 400mg every 12 hours, maraviroc 300mg every 12 hours (AM doses only on Day 14)
- Raltegravir (Reference): 400 mg every 12 hours on Study Days 1-3 Followed by washout on Study Days 4-5
Arm/Group | Maraviroc + Raltegravir (Test) | Raltegravir (Reference)
Number analyzed (Participants) | 17 | 18
ng.hr/mL | 6287.5 (3979.30) | 9122.4 (5311.34)
Statistical Analysis 1: Comparison: Maraviroc + Raltegravir (Test) vs Raltegravir (Reference); For raltegravir, a sample size of 18 subjects provided 90% CIs for the difference between treatments of raltegravir (±0.205) on the natural log scale for AUCτ, with 90% coverage probability; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio (percent) = 63.25, 90% CI [44.27 to 90.39] — Ratio (percent) (Test/Reference) of Adjusted Geometric Means

4. Other Pre Specified Outcome: Maraviroc Pharmacokinetic (PK) Parameter: 12-Hour Trough Concentration (C12)
Description: Effect of raltegravir on pharmacokinetics of maraviroc (comparison of C12 of raltegravir co-administered with maraviroc (Test) versus maraviroc administered alone (Reference)). Pharmacokinetics were assessed on Day 11 (maraviroc) and Day 14 (maraviroc and raltegravir). C12 is the 12-hour trough concentration.
Time Frame: Days 11 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Maraviroc + Raltegravir (Test) | Maraviroc (Reference)
Number analyzed (Participants) | 17 | 17
ng/mL | 48.34 (13.70) | 53.36 (14.03)
Statistical Analysis 1: Comparison: Maraviroc + Raltegravir (Test) vs Maraviroc (Reference); The alternate hypothesis of bioequivalence is that there is no difference between treatment groups; Test type: Superiority or Other; Mixed Models Analysis; Natural log transformed C12 was analyzed using a mixed effect model with treatment as a fixed effect and subject as a random effect; Ratio (percent) = 90.33, 90% CI [85.28 to 95.68] — Ratio (percent) (Test/Reference) of Adjusted Geometric Means

5. Primary Outcome: Raltegravir Pharmacokinetics (PK) Parameter: Maximum Concentration (Cmax)
Description: Effect of maraviroc on pharmacokinetics of raltegravir (comparison of Cmax of raltegravir co-administered with maraviroc (Test) versus raltegravir administered alone (Reference)). Pharmacokinetics assessed on Day 3 (raltegravir) and Day 14 (maraviroc and raltegravir). Cmax is the maximum plasma concentration.
Time Frame: Days 3 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Maraviroc + Raltegravir (Test) | Raltegravir (Reference)
Number analyzed (Participants) | 17 | 18
ng/mL | 2169.6 (1570.58) | 3026.6 (2030.15)
Statistical Analysis 1: Comparison: Maraviroc + Raltegravir (Test) vs Raltegravir (Reference); For raltegravir, a sample size of 18 subjects provided 90% CIs for the difference between treatments of raltegravir (±0.293) on the natural log scale for Cmax, with 90% coverage probability; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Ratio (percent) = 66.77, 90% CI [41.22 to 108.15] — Ratio (percent) (Test/Reference) of Adjusted Geometric Means

6. Other Pre Specified Outcome: Raltegravir Pharmacokinetics (PK) Parameter: 12-Hour Trough Concentration (C12)
Description: Effect of maraviroc on pharmacokinetics of raltegravir (comparison of C12 of raltegravir co-administered with maraviroc (Test) vs. raltegravir administered alone (Reference)). Pharmacokinetics were assessed on Day 3 (raltegravir) and Day 14 (maraviroc and raltegravir). C12 is the 12-hour trough concentration.
Time Frame: Days 3 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Maraviroc + Raltegravir (Test) | Raltegravir (Reference)
Number analyzed (Participants) | 17 | 18
ng/mL | 51.16 (22.64) | 73.69 (36.21)
Statistical Analysis 1: Comparison: Maraviroc + Raltegravir (Test) vs Raltegravir (Reference); Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 4, analysis 1]; ratio (percent) = 72.42, 90% CI [57.82 to 90.71] — Ratio (percent) (Test/Reference) of Adjusted Geometric Means

ADVERSE EVENTS:
Groups:
- Maraviroc: 300 milligrams (mg) every 12 hours on Study Days 6-11
- Maraviroc + Raltegravir: On Study Days 12-14: Raltegravir 400 milligrams (mg) every 12 hours, maraviroc 300 mg every 12 hours (AM doses only on Day 14)
- Raltegravir: 400 milligrams (mg) every 12 hours on Study Days 1-3 Followed by washout on Study Days 4-5
Arm/Group | Maraviroc | Maraviroc + Raltegravir | Raltegravir
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 4 | 4 | 3
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Maraviroc | Maraviroc + Raltegravir | Raltegravir
Constipation (Gastrointestinal disorders) | 1/18 | 0/17 | 0/18
Dyspepsia (Gastrointestinal disorders) | 0/18 | 1/17 | 0/18
Folliculitis (Infections and infestations) | 1/18 | 0/17 | 1/18
Back pain (Musculoskeletal and connective tissue disorders) | 0/18 | 1/17 | 0/18
Headache (Nervous system disorders) | 0/18 | 1/17 | 2/18
Peripheral neurophathy (Nervous system disorders) | 1/18 | 1/17 | 1/18
Somnolence (Nervous system disorders) | 1/18 | 1/17 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.